CLINICAL TRIAL: NCT00853515
Title: A Randomized-controlled Trial of a Targeted Approach to Fluid Resuscitation in Acute Pancreatitis
Brief Title: Goal-directed Fluid Resuscitation in Acute Pancreatitis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: interim analysis incidence primary endpoint lower than anticipated. Sigicant finding based on secondary endpoint.
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Bechien Wu, MD, MPH, Bechien Wu, M.D., M.P.H., Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-P-001757
Record Dates: First submitted 2009-02-27; First posted 2009-03-02 (Estimated); Last update posted 2016-12-09 (Estimated); Status verified 2016-12

CONDITIONS: Acute Pancreatitis
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): Goal-directed fluid resuscitation with lactated Ringer's solution
  Interventions: Other: Goal-directed fluid resuscitation
- 2 (Experimental): Goal-directed fluid resuscitation with normal saline
  Interventions: Other: Goal-directed fluid resuscitation
- 3 (No Intervention): Standard fluid resuscitation with lactated Ringer's solution
- 4 (No Intervention): Standard fluid resuscitation with normal saline

INTERVENTIONS:
Other: Goal-directed fluid resuscitation — Targeted, weight-based fluid resuscitation
  Arms: 1; 2

SUMMARY:
Vigorous fluid resuscitation is currently believed to play a key role in reducing complications associated with acute pancreatitis. However, aggressive fluid replacement can be associated with complications such as pulmonary fluid sequestration. The purpose of this study is to evaluate alternative approaches to early fluid resuscitation for patients with acute pancreatitis.

DETAILED DESCRIPTION:
Primary Aim: Evaluate the impact of a goal-directed fluid resuscitation protocol compared to standard fluid resuscitation on systemic inflammation in patients with acute pancreatitis.

Secondary Aim: Evaluate the impact of resuscitation with Lactated Ringer's compared to normal saline on systemic inflammation in acute pancreatitis.

ELIGIBILITY:
Inclusion Criteria:

* acute pancreatitis diagnosed by at least 2 criteria
* adult patients at least 18 years of age

Exclusion Criteria:

* history of severe cardiovascular, respiratory, renal, hepatic or hematologic/immunologic disease
* concurrent metabolic or physiologic derangement requiring specific fluid management
* pregnancy
* patients transferred from acute care hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-03; Primary Completion 2010-02 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Prevalence (point prevalence) of the systemic inflammatory response syndrome (SIRS) at 24 hours | first 24 hours of hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Bechien U. Wu, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States